CLINICAL TRIAL: NCT05439109
Title: To Evaluate the Appropriate Depth of Endotracheal Tube Placement Guided by Topographical Landmarks
Brief Title: Correct Endotracheal Tube Placement Using Topographical Landmarks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Dr. Amit Kumar Mittal, Principal Investigator, Rajiv Gandhi Cancer Institute & Research Center, India
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RES/SCM/35/2019/68
Record Dates: First submitted 2022-06-21; First posted 2022-06-30 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Intubation, Intratracheal; Anatomic Landmarks
Keywords: Endotracheal tube placement; Topographical landmarks of trachea

STUDY DESIGN:
Intervention Model Description: All enrolled patients will be intubated by either topographical landmarks of individual tracheal dimensions or by the conventional intubation guide method.
Who Masked: Participant, Outcomes Assessor
Masking Description: The primary investigator will provide the information regarding the portion of endotracheal to be kept below the vocal cords to the care provider after measuring the dimensions of the trachea topographically. After tube placement, the tube tip to carina distance will be measured in both topographical and intubation guide mark technique.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Topographical landmark technique (Experimental): Surface anatomic landmarks of an individual's trachea will be measured from the mid-thyroid level (corresponds to vocal cords) to manubriosternal joint (corresponds to carina) in the sagittal plane to estimate tracheal length. Three centimeters will be deducted from the estimated tracheal length to provide the length of the endotracheal tube from the tube tip to be inserted inside the trachea.
  Interventions: Device: Topographical landmark technique of endotracheal tube placement
- Intubation guide mark technique (Active Comparator): Already established and commonly practiced technique, in this technique, the guide mark present above the proximal end of the endotracheal tube cuff will be placed just beyond the vocal cords.
  Interventions: Device: Intubation guide mark technique of endotracheal tube placement

INTERVENTIONS:
Device: Topographical landmark technique of endotracheal tube placement — An endotracheal tube will be placed inside the trachea after measuring the individual's estimated tracheal dimensions.
  Arms: Topographical landmark technique
Device: Intubation guide mark technique of endotracheal tube placement — An endotracheal tube will be placed in this group by using the intubation guide mark.
  Arms: Intubation guide mark technique

SUMMARY:
An optimal endotracheal tube depth is ideally required for preventing the complications associated with mal-positioning of the endotracheal tube. The topographical technique of tube placement considering the individual's morphometric dimensions could help to provide optimal tube placement. hence, to evaluate the efficacy of the topographical technique in providing the optimal tube placement this study will be conducted.

DETAILED DESCRIPTION:
The trachea is a dynamic organ and its length varies by various static and dynamic factors leading to changing the tracheal length and variable endotracheal tube tip to carina (Ti-Ca) distance. Hence, upholding optimal Ti-Ca distance during changing tracheal length is of utmost importance to prevent complications associated with endotracheal tube (ETT) mal-positioning. When the length of ETT, which is to be inserted inside the trachea, is calculated as per an individual's tracheal morphometric dimensions, the appropriate depth of placement could be achieved and tube malpositioning can be prevented. In the topographical landmark technique, an individual tracheal length is estimated by measuring the various distance from mid-thyroid level (corresponds to vocal cords) to manubriosternal joint (corresponds to carina) in the sagittal plane. After estimating the tracheal length, tip to carina distance of 3cm was deducted from the estimated length of the trachea to provide the distance of the endotracheal tube to be kept beyond the vocal cords. Hence, the investigators planned this study to find the "utility and reliability" of the topographical landmark technique compared to the conventional intubation guide mark technique in providing the appropriate depth of endotracheal tube placement.

ELIGIBILITY:
Inclusion Criteria:

* • Age group of 18-75 years

  * ASA physical status I-III patients
  * Oral intubation for general anesthesia

Exclusion Criteria:

* • Patient with upper airway fibrosis

  * Tracheal stenosis or tracheal surgeries
  * Previous head and neck surgeries
  * Contracture neck or irradiated neck
  * Large neck swelling distorting or deviating the trachea
  * Laryngeal or tracheal tumor
  * Intubations requiring flexo-metallic tubes
  * Patient refusal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Endotracheal tube position inside the trachea | through study completion approximately at six months
  Tip to carina distance will be measured by fiber optic bronchoscopy to classify the optimal or suboptimal tube placements in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Amit K Mittal, M.D, Principal Investigator — Senior Consultant, Department of Anesthesiology, Rajiv Gandhi Cancer Institute and Research centre
Locations (1):
- Amit, Rohini, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided
If necessary IPD data can be disclosed after patients approval.